CLINICAL TRIAL: NCT03236350
Title: The Effect of Remote Ischaemic Conditioning on Blood Pressure Control in Patients With Chronic Kidney Disease - the ERIC-BP-CKD Trial
Brief Title: Remote Ischaemic Conditioning on Blood Pressure Control in Chronic Kidney Disease Patients
Acronym: ERIC-BP-CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHF/CTG059/2016
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Diseases; Hypertension; Cardiovascular Diseases
Keywords: Chronic Kidney Disease; Hypertension; Cardiovascular Disease; Central Aortic Systolic Pressure; Proteinuria; Remote Ischemic Conditioning; Left Ventricular Hypertrophy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Cardiovascular Diseases; Proteinuria; Hypertrophy, Left Ventricular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRIC Treatment (Experimental): An autoRIC® Device will be placed on the upper arm daily to complete the preset protocol and will be repeated daily for 28 days.
  Interventions: Device: Active autoRIC® (CRIC Treatment)
- Sham Control (Sham Comparator): An autoRIC® Device visually identical to that used in the CRIC protocol will be placed on the upper arm daily to complete the preset protocol and will be repeated daily for 28 days.
  Interventions: Device: Sham Control autoRIC® (Sham Control)

INTERVENTIONS:
Device: Active autoRIC® (CRIC Treatment) — The active autoRIC® Device is programmed to go through a preset protocol of inflation and deflation cycles every session. The sessions will be repeated daily for 28 days.
  Arms: CRIC Treatment
Device: Sham Control autoRIC® (Sham Control) — The Sham Control autoRIC® Device is visually identical to the active autoRIC® Device but the simulated protocol applied comprises of vibrations of the device but no inflation of the cuff every session. The sham device provides the same sound and vibration as that of the pump inflating and the same LED indicators on the Active Unit. The sessions will be repeated daily for 28 days.
  Arms: Sham Control

SUMMARY:
Chronic kidney disease (CKD) is one of the leading causes of death and disability in Singapore and worldwide. Hypertension is commonly inadequately controlled in patients with CKD and this is associated with CKD progression and cardiovascular complications. Daily episodes of Remote ischaemic conditioning (termed chronic RIC or CRIC) using transient limb ischaemia/reperfusion applied for 1 to 12 months have been shown to lower systemic blood pressure (SBP), prevent stroke and reduce post-myocardial infarction left ventricular (LV) remodelling in experimental and clinical studies. In the ERIC-BP-CKD feasibility and efficacy study, we hypothesise that CRIC administered for 28 days will lower systemic blood pressure and improve blood pressure control in patients with CKD and hypertension.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is one of the leading causes of death and disability in Singapore and worldwide. CKD patients often suffer with inadequately controlled hypertension, the presence of which is associated with cardiovascular complications such as left ventricular (LV) hypertrophy, cardiac failure, and stroke. As such, novel treatments are required to improve blood pressure control in order to improve health outcomes in CKD patients.

Remote ischaemic conditioning (RIC) using transient limb ischaemia/reperfusion has been shown to protect the kidney and microvasculature in experimental and clinical studies, and daily episodes of RIC (termed chronic RIC or CRIC) applied for 1 to 12 months have been shown to lower systemic blood pressure (SBP), prevent stroke and reduce post-myocardial infarction left ventricular (LV) remodelling in experimental and clinical studies. Whether CRIC can reduce SBP in hypertensive patients with CKD is not known. In the ERIC-BP-CKD feasibility and efficacy study, we hypothesise that CRIC administered for 28 days will lower systemic blood pressure and improve blood pressure control in patients with CKD and hypertension.

In this study, subjects will be randomised in a 1:1 ratio to receive therapy from either the active autoRIC® Device or identical sham autoRIC® Device.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Aged 21 years and older
3. CKD (all stages 1-4)
4. On treatment for hypertension and automated office BP (AOBP) ≥ 140mmHg (this will be determined by an automated oscillometric BP device)

Exclusion Criteria:

1. Patients with polycystic kidney disease
2. Atrial fibrillation
3. Patients on long-acting sulphonylureas (eg glibenclamide) or nicorandil (as these medications may interfere with the protective effect of CRIC).
4. Patients recruited into another study which may impact on this study.
5. Symptomatic peripheral arterial disease affecting the upper limbs (given nature of upper-limb CRIC protocol).
6. Renal transplant / Dialysis patients
7. Pregnant patients
8. Patients on any anti-coagulant medications (e.g. Warfarin)
9. For echo sub-study only: Prior myocardial infarction, BMI > 30kg/m2, known severe acrdiac valve disease, known severely impaired LVEF <35%

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline and 28 days
  Difference in change in systolic blood pressure (measured by automated office blood pressure recording) from baseline to after 28 days between CRIC versus sham control therapy.

SECONDARY OUTCOMES:
Number of antihypertensive medications | Baseline and 28 days
  Reduction in number of medications required for treating hypertension
Central aortic systolic pressure | Baseline and 28 days
  Central aortic systolic pressure (measured by assessing the arterial waveform after 28 days of CRIC or sham control therapy).
Arterial pulse waveform | Baseline and 28 days
  The arterial pulse waveform (measured after 28 days of CRIC or sham control therapy).
LV systolic and diastolic function | Baseline and 28 days
  Change in LV systolic and diastolic function assessed by echocardiography from baseline following 28 days of CRIC or sham control therapy (subset of 20 patients).
LV wall thickness | Baseline and 28 days
  Change in LV wall thickness assessed by echocardiography from baseline following 28 days of CRIC or sham control therapy (subset of 20 patients).
Spot Urine Protein-Creatinine Ratio | Baseline and 28 days
  Change in Proteinuria assessed by Spot Urine Protein-Creatinine Ratio from baseline after 28 days of CRIC or sham control therapy.
Serum creatinine and eGFR | Baseline and 28 days
  Change in Renal function (assessed by serum creatinine and eGFR from baseline to after 28 days of CRIC or sham control therapy).
Blood biomarkers for CKD and inflammation | Baseline and 28 days
  CRP, IL-6, PAI-1, sCD40 ligand, and TNF-alpha will be measured for CKD and inflammation following 28 days of CRIC or sham control therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Choo, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Result] Luca MC, Liuni A, McLaughlin K, Gori T, Parker JD. Daily ischemic preconditioning provides sustained protection from ischemia-reperfusion induced endothelial dysfunction: a human study. J Am Heart Assoc. 2013 Feb 22;2(1):e000075. doi: 10.1161/JAHA.112.000075. PMID 23525419